CLINICAL TRIAL: NCT03163550
Title: A Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, Food Effect, and the Drug-Drug Interaction Potential of Oral ACHN-383 and ACHN-789 in Healthy Subjects
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, Food Effect, and Drug-Drug Interaction Potential of ACHN-383 and ACHN-789
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achaogen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACHN-172-001
Record Dates: First submitted 2017-05-15; First posted 2017-05-23 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Healthy volunteers
  Interventions: Drug: ACHN-383; Drug: ACHN-789; Drug: Placebo
- Cohort 2 (Experimental): Healthy volunteers
  Interventions: Drug: ACHN-383; Drug: ACHN-789; Drug: Placebo
- Cohort 3 (Experimental): Healthy volunteers
  Interventions: Drug: ACHN-383; Drug: ACHN-789; Drug: Placebo
- Cohort 4 (Experimental): Healthy volunteers
  Interventions: Drug: ACHN-383; Drug: ACHN-789; Drug: Placebo
- Cohort 5 (Experimental): Healthy volunteers
  Interventions: Drug: ACHN-383; Drug: ACHN-789; Drug: Placebo

INTERVENTIONS:
Drug: ACHN-383 — Oral dose
Drug: ACHN-789 — Oral dose
Drug: Placebo — Oral dose

SUMMARY:
This Phase 1 clinical study is a double-blind, randomized, placebo-controlled, parallel group study to assess the safety, tolerability, pharmacokinetics (PK), food effect, and drug interaction potential of ACHN-383 and ACHN-789 co-administered orally as separate capsules in healthy subjects

ELIGIBILITY:
Key Inclusion Criteria:

* Females of child-bearing potential must not be breast feeding, must have a negative serum pregnancy test, and must use a highly effective method of contraception or be abstinent from sexual activity prior to the first dose of study, during the study and for a specified period following the last dose of study drug
* Males must be willing to use a condom for the duration of the study and for a specified period following the study, unless surgically sterile. In addition, their female partner must use a highly effective method of contraception, for the same period of time, unless surgically sterile
* Body mass index (BMI) of ≥19 kg/m^2 to ≤32 kg/m^2 and weight ≥50 kg to ≤125 kg
* Normal renal function as determined by creatinine clearance (CLcr) rate

Key Exclusion Criteria:

* Pregnant women
* History of any hepatic or biliary disorder or disease
* Any condition that could possibly affect oral drug absorption
* Unstable cardiovascular disease
* Uncontrolled hypertension, asthma, diabetes, thyroid disease, or seizure disorder
* HIV positive
* Active malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in clinical laboratory values (CBC, serum chemistry, urine analysis, AST, ALT, ALP, serum bilirubin) | 26 days
Changes from baseline in vital signs (temperature, pulse, respiration, blood pressure) | 26 days
Incidence and severity of adverse events | 26 days
Changes from baseline in the QTcF interval | 19 days

SECONDARY OUTCOMES:
PK parameter: Maximum peak observed concentration (Cmax) after single-dose administration of ACHN-789 | 1 day
PK parameter: Maximum peak observed concentration (Cmax) after single-dose administration of ACHN-383 | 3 days
PK parameter: Time to maximum concentration (Tmax) after single-dose administration of ACHN-789 | 1 day
PK parameter: Time to maximum concentration (Tmax) after single-dose administration of ACHN-383 | 3 days
PK parameter: Area under the concentration-time curve (AUC) after single-dose administration of ACHN-789 | 1 day
PK parameter: Area under the concentration-time curve (AUC) after single-dose administration of ACHN-383 | 3 days
PK parameter: Half-life (t1/2) after single-dose administration of ACHN-789 | 1 day
PK parameter: Half-life (t1/2) after single-dose administration of ACHN-383 | 3 days
PK parameter: Apparent systemic clearance (CL/F) after single-dose administration of ACHN-789 | 1 day
PK parameter: Apparent systemic clearance (CL/F) after single-dose administration of ACHN-383 | 3 days
PK parameter: Apparent volume of distribution (Vz/F) after single-dose administration of ACHN-789 | 1 day
PK parameter: Apparent volume of distribution (Vz/F) after single-dose administration of ACHN-383 | 3 days
PK parameter: Amount excreted in urine (Ae) after single-dose administration of ACHN-789 | 1 day
PK parameter: Amount excreted in urine (Ae) after single-dose administration of ACHN-383 | 3 days
PK parameter: Renal clearance (CLr) after single-dose administration of ACHN-789 | 1 day
PK parameter: Renal clearance (CLr) after single-dose administration of ACHN-383 | 3 days
PK parameter: Cmax after single-dose administration of ACHN-383 and ACHN-789 given concurrently | 1 day
PK parameter: Cmax after single-dose administration of ACHN-383 and ACHN-789 given concurrently | 5 days
PK parameter: Tmax after single-dose administration of ACHN-383 and ACHN-789 given concurrently | 1 day
PK parameter: Tmax after single-dose administration of ACHN-383 and ACHN-789 given concurrently | 5 days
PK parameter: AUC after single-dose administration of ACHN-383 and ACHN-789 given concurrently | 1 day
PK parameter: AUC after single-dose administration of ACHN-383 and ACHN-789 given concurrently | 5 days
PK parameter: t1/2 after single-dose administration of ACHN-383 and ACHN-789 given concurrently | 1 day
PK parameter: t1/2 after single-dose administration of ACHN-383 and ACHN-789 given concurrently | 5 days
PK parameter: CL/F after single-dose administration of ACHN-383 and ACHN-789 given concurrently | 1 day
PK parameter: CL/F after single-dose administration of ACHN-383 and ACHN-789 given concurrently | 5 days
PK parameter: Vz/F after single-dose administration of ACHN-383 and ACHN-789 given concurrently | 1 day
PK parameter: Vz/F after single-dose administration of ACHN-383 and ACHN-789 given concurrently | 5 days
PK parameter: Ae after single-dose administration of ACHN-383 and ACHN-789 given concurrently | 1 day
PK parameter: Ae after single-dose administration of ACHN-383 and ACHN-789 given concurrently | 5 days
PK parameter: CLr after single-dose administration of ACHN-383 and ACHN-789 given concurrently | 1 day
PK parameter: CLr after single-dose administration of ACHN-383 and ACHN-789 given concurrently | 5 days
PK parameter: Cmax after single-dose administration of ACHN-383 and ACHN-789 given concurrently 30 minutes after a high-fat, high-calorie meal | 6 days
PK parameter: Tmax after single-dose administration of ACHN-383 and ACHN-789 given concurrently 30 minutes after a high-fat, high-calorie meal | 6 days
PK parameter: AUC after single-dose administration of ACHN-383 and ACHN-789 given concurrently 30 minutes after a high-fat, high-calorie meal | 6 days
PK parameter: t1/2 after single-dose administration of ACHN-383 and ACHN-789 given concurrently 30 minutes after a high-fat, high-calorie meal | 6 days
PK parameter: CL/F after single-dose administration of ACHN-383 and ACHN-789 given concurrently 30 minutes after a high-fat, high-calorie meal | 6 days
PK parameter: Vz/F after single-dose administration of ACHN-383 and ACHN-789 given concurrently 30 minutes after a high-fat, high-calorie meal | 6 days
PK parameter: Ae after single-dose administration of ACHN-383 and ACHN-789 given concurrently 30 minutes after a high-fat, high-calorie meal | 6 days
PK parameter: CLr after single-dose administration of ACHN-383 and ACHN-789 given concurrently 30 minutes after a high-fat, high-calorie meal | 6 days
PK parameter: Cmax after multiple-dose administration of ACHN-383 and ACHN-789 given concurrently | 19 days
PK parameter: Cmin after multiple-dose administration of ACHN-383 and ACHN-789 given concurrently | 19 days
PK parameter: Tmax after multiple-dose administration of ACHN-383 and ACHN-789 given concurrently | 19 days
PK parameter: AUC after multiple-dose administration of ACHN-383 and ACHN-789 given concurrently | 19 days
PK parameter: t1/2 after multiple-dose administration of ACHN-383 and ACHN-789 given concurrently | 19 days
PK parameter: CL/F after multiple-dose administration of ACHN-383 and ACHN-789 given concurrently | 19 days
PK parameter: Vz/F after multiple-dose administration of ACHN-383 and ACHN-789 given concurrently | 19 days
PK parameter: Ae after multiple-dose administration of ACHN-383 and ACHN-789 given concurrently | 19 days
PK parameter: CLr after multiple-dose administration of ACHN-383 and ACHN-789 given concurrently | 19 days
Urine concentrations of ACHN-789 after single dose administration | 1 day
Urine concentrations of ACHN-383 after single-dose administration | 3 days
Urine concentrations of ACHN-383 and ACHN-789 after single-dose administration given concurrently | 1 day
Urine concentrations of ACHN-383 and ACHN-789 after single-dose administration given concurrently | 5 days
Urine concentrations of ACHN-383 and ACHN-789 after multiple-dose administration given concurrently | 19 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Cloutier, PharmD, Study Director — Achaogen, Inc.
Locations (1):
- Clinical Site, Perth, Australia